CLINICAL TRIAL: NCT05560763
Title: FlowTriever Pulmonary Embolectomy Clinical Study - FlowTriever2
Brief Title: FlowTriever2 Pulmonary Embolectomy Clinical Study
Acronym: FLARE-FT2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inari Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-001
Record Dates: First submitted 2022-09-21; First posted 2022-09-29 (Actual); Results first posted 2025-09-23 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- All Subjects (Experimental): All participants who were treated with the FlowTriever System and FlowTriever2 Catheter.
  Interventions: Device: FlowTriever2 Catheter

INTERVENTIONS:
Device: FlowTriever2 Catheter — The FlowTriever2 Catheter is utilized for the treatment of Pulmonary Embolism via mechanical thrombectomy of thrombus in the pulmonary arteries.

SUMMARY:
The FLARE-FT2 confirmatory study is a prospective, single-arm, multicenter study of the FlowTriever2 Catheter for mechanical thrombectomy of pulmonary embolism (PE).

DETAILED DESCRIPTION:
The study is a prospective, single-arm, multicenter study to evaluate the safety and effectiveness of the FlowTriever2 Catheter for mechanical thrombectomy in patients eligible for endovascular treatment of acute pulmonary embolism (PE). The subjects who meet the inclusion/exclusion criteria will be enrolled in the study. The enrollment period is over a period of approximately 12 months. All study subjects actively participate through the 30-day visit (-5 / +15 days) following treatment. Study participation includes screening, baseline, treatment, 48-hour visit, and 30-day follow-up. The study population consists of subjects that have an acute PE. Subject eligibility is determined based on data available to the Investigator at the time of enrollment. Subjects must meet all inclusion and no exclusion criteria to be eligible for the study. All subjects that complete the procedure and the follow-ups are included in the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical signs and symptoms consistent with acute PE
* PE symptom duration ≤ 14 days
* CTA evidence of proximal PE (filling defect in at least one main or lobar pulmonary artery)
* RV/LV ratio of ≥ 0.9 (NOTE: Enrollment qualification assessment based on Investigator's interpretation of RV/LV ratio)
* Systolic blood pressure ≥ 90 mmHg (initial SBP may be ≥ 80 mmHg if the pressure recovers to ≥ 90 mmHg with fluids)
* Stable heart rate < 130 BPM prior to procedure
* Patient is deemed medically eligible for interventional procedure(s), per institutional guidelines and/or clinical judgment.
* FlowTriever2 Catheter enters the vasculature

Exclusion Criteria:

* Thrombolytic use within 30 days of baseline CTA
* Pulmonary hypertension with peak pulmonary artery pressure > 70 mmHg by right heart catheterization
* Vasopressor requirement after fluids to keep pressure ≥ 90 mmHg
* FiO2 requirement > 40% or > 6 LPM to keep oxygen saturation > 90%
* Hematocrit < 28% (NOTE: hematocrit required within 6 hours of index procedure)
* Platelets < 100,000/μL
* Serum creatinine > 1.8 mg/dL
* INR > 3
* Major trauma Injury Severity Score (ISS) > 15
* Presence of intracardiac lead in the right ventricle or right atrium placed within 6 months
* Cardiovascular or pulmonary surgery within last 7 days
* Actively progressing cancer
* Known bleeding diathesis or coagulation disorder
* Left bundle branch block
* History of severe or chronic pulmonary arterial hypertension
* History of chronic left heart disease with left ventricular ejection fraction ≤ 30%
* History of uncompensated heart failure
* History of underlying lung disease that is oxygen dependent
* History of chest irradiation
* History of heparin-induced thrombocytopenia (HIT) Any contraindication to systemic or therapeutic doses heparin or anticoagulants
* Known anaphylactic reaction to radiographic contrast agents that cannot be pretreated
* Imaging evidence or other evidence that suggests, in the opinion of the Investigator, the Subject is not appropriate for mechanical thrombectomy intervention (e.g., inability to navigate to target location, predominately chronic clot, or non-clot embolus)
* Life expectancy of < 90 days, as determined by Investigator
* Female who is pregnant or nursing
* Current participation in another investigational drug or device treatment study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-02-14 (Actual); Primary Completion 2024-09-09 (Actual); Study Completion 2024-09-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Carondelet St. Joseph's Hospital, Tucson, Arizona
  - Yale University, New Haven, Connecticut
  - Memorial Health University Medical Center, Savannah, Georgia
  - Baptist Health, Louisville, Kentucky
  - Virtua Health, Camden, New Jersey
  - Oklahoma Heart Institute, Tulsa, Oklahoma
  - University of Tennessee Medical Center, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects presenting to the hospital/emergency department with a pulmonary embolism (PE) and meeting all eligibility requirements for enrollment in the FLARE-FT2 study.
Groups:
- All Subjects: All participants who were treated with the FlowTriever System and FlowTriever2 Catheter for mechanical thrombectomy of PE.
Period: Overall Study
Arm/Group | All Subjects
Started | 50 (50 subjects completed FlowTriever procedures; 8 subjects were later discovered to violate the exclusion criteria per protocol and excluded from the Enrollment Population.)
Enrollment Population (Enrollment Population includes all patients who met the inclusion/exclusion criteria and in whom the FlowTriever2 Catheter is inserted into the vasculature.) | 42
Intent-to-Treat Population (Intent-to-Treat Population includes all enrolled subjects who met the inclusion/exclusion criteria and in whom the procedure was attempted, and the FlowTriever2 Catheter was deployed, whether successful or not.) | 42
Modified Intent-to-Treat Population (Modified Intent-to-Treat Population includes all subjects in the Intent-to-Treat Population who have no thrombolytics administered during the procedure.) | 42
Full Analysis Set Population (Full Analysis Set Population includes all subjects in the Modified Intent-to-Treat Population that have successfully received the procedure and have completed the 48-hour post-procedure follow-up (+36 hours or discharge, whichever comes first) per study protocol.) | 42
Completed Cases Population (Completed Cases Population includes all subjects in the Modified Intent-to-Treat Population that have successfully received the procedure and have completed all follow-up visits.) | 38
Completed | 46
Not Completed | 4
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | All Subjects
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (12.08)
Age, Continuous [Median (Full Range); unit: years] | 63 [27 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 46
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 37
  More than one race | 0
  Unknown or Not Reported | 1
Height (m) [Median (Full Range); unit: m] | 1.75 [1.5 to 1.9]
Weight (kg) [Median (Full Range); unit: kg] | 99.9 [47.2 to 172.4]
BMI (kg/m^2) [Median (Full Range); unit: kg/m^2] | 33.2 [17.6 to 53.0]
Tobacco Use [Count of Participants; unit: Participants]
  Current | 12
  Past | 12
  Never | 26
Prior Pulmonary Embolism (PE) [Count of Participants; unit: Participants]
  Yes | 8
  No | 42
Prior deep venous thrombosis (DVT) [Count of Participants; unit: Participants]
  Yes | 14
  No | 36
History of pulmonary hypertension [Count of Participants; unit: Participants]
  Yes | 2
  No | 48
History of systemic hypertension [Count of Participants; unit: Participants]
  Yes | 28
  No | 22
History of coronary artery disease (CAD) [Count of Participants; unit: Participants]
  Yes | 4
  No | 46
History of congestive heart failure (CHF) [Count of Participants; unit: Participants]
  Yes | 3
  No | 47
History of coronary artery bypass graft (CABG) [Count of Participants; unit: Participants]
  Yes | 0
  No | 50
History of chronic obstructive pulmonary disease (COPD) [Count of Participants; unit: Participants]
  Yes | 4
  No | 46
History of myocardial infarction (MI) [Count of Participants; unit: Participants]
  Yes | 2
  No | 48
Patent foramen ovale (PFO) / shunt [Count of Participants; unit: Participants]
  Yes | 1
  No | 49
Prior cerebrovascular accident (prior stroke/transient ischemic attack (TIA)) [Count of Participants; unit: Participants]
  Yes | 1
  No | 49
Hypercoagulable state [Count of Participants; unit: Participants]
  Yes | 0
  No | 50
History of cancer [Count of Participants; unit: Participants]
  Yes | 7
  No | 43
Active Cancer [Count of Participants; unit: Participants] — Population: This analysis is only applied to subjects that have a history of cancer (7).
  Participants
    number analyzed (Participants) | 7
    Yes | 0
    No | 7
History of renal disease (chronic renal insufficiency) [Count of Participants; unit: Participants]
  Yes | 3
  No | 47
On dialysis [Count of Participants; unit: Participants] — Population: This analysis is only applied to subjects that have a history of renal disease (chronic renal insufficiency) (3).
  Participants
    number analyzed (Participants) | 3
    Yes | 0
    No | 3
Recent surgery (within 30 days) [Count of Participants; unit: Participants]
  Yes | 6
  No | 44
Recent surgery type [Count of Participants; unit: Participants] — Population: This analysis is only applied to subjects that have had recent surgery (within the last 30 days) (6).
  Participants
    number analyzed (Participants) | 6
    Orthopedic | 2
    Neurological | 1
    Abdomen | 1
    Other | 2
Recent trauma (within 30 days) [Count of Participants; unit: Participants]
  Yes | 1
  No | 49
Thrombolytic contraindication [Count of Participants; unit: Participants]
  None | 48
  Relative | 1
  Absolute | 1
Relative thrombolytic contraindication [Number; unit: Condition applies to subject] — Population: This analysis is only applied to subjects that have relative thrombolytic contraindication (1).
  Condition applies to subject
    Oral anticoagulation except for aspirin: number analyzed (Participants) | 1
    Oral anticoagulation except for aspirin | 1
    Therapeutic LMWH within 24 hours: number analyzed (Participants) | 1
    Therapeutic LMWH within 24 hours | 1
Absolute thrombolytic contraindication with recent intracranial/spinal surgery or head trauma [Count of Participants; unit: Participants] — Population: This analysis is only applied to subjects that have an absolute thrombolytic contraindication (1).
  Participants
    number analyzed (Participants) | 1
    (all) | 1
History of diabetes [Count of Participants; unit: Participants]
  Yes | 14
  No | 36
Diabetes type [Count of Participants; unit: Participants] — Population: This analysis is only applied to subjects that have diabetes (14).
  Participants
    number analyzed (Participants) | 14
    Diabetes mellitus type 1 | 1
    Diabetes mellitus type 2 | 13
Current COVID-19 status [Count of Participants; unit: Participants]
  COVID-19 positive | 1
  COVID-19 negative | 12
  COVID-19 status unknown | 37
Prior COVID-19 infection [Count of Participants; unit: Participants]
  Previously recovered | 6
  Prior infection unknown | 33
  Not applicable | 11

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Endpoint (Composite): Incidence of Adjudicated Serious Adverse Events (SAE)
Description: Incidence of adjudicated Serious Adverse Events (SAE), which is a composite of:
  * Mortality through 48 hours after the index procedure related to FlowTriever2 Catheter
  * Major bleeding through 48 hours after the index procedure related to FlowTriever2 Catheter
  * Intra-procedural device or procedure-related adverse events, including:
    * Clinical deterioration defined by hemodynamic or respiratory worsening
    * Pulmonary vascular injury related to FlowTriever2 Catheter
    * Cardiac injury related to FlowTriever2 Catheter
Time Frame: Device-related mortality and device-related major bleeding components assessed through 48 hours after index procedure. Intra-procedural device or procedure-related AE component assessed until index procedure completion (index procedure: approx. 50 mins).
Measure: Count of Participants; unit: Participants
Arm/Group | All Subjects
Number analyzed (Participants) | 50
Participants
  Yes | 0
  No | 50

2. Primary Outcome: Primary Effectiveness Endpoint: Change in Mean Pulmonary Arterial Pressure (mmHg)
Description: Change in mean pulmonary arterial pressure measured via right heart catheterization at the beginning of the treatment procedure and at the end of the treatment procedure.
Time Frame: Intraprocedural (at beginning and end of treatment procedure (index procedure: approximately 50 minutes))
Measure: Median (Full Range); unit: mmHg
Arm/Group | All Subjects
Number analyzed (Participants) | 50
mmHg | -5.50 [-29.0 to 15.0]

3. Secondary Outcome: Secondary Safety Endpoint: Number of Patient Mortalities
Description: Number of adjudicated all-cause mortalities through the 30-day visit (visit window = 30 days from procedure -5 / +15 days)
Time Frame: 30 days post procedure (-5 / +15 days)
Measure: Count of Participants; unit: Participants
Arm/Group | All Subjects
Number analyzed (Participants) | 50
Participants
  Yes | 0
  No | 46
  Withdrawn | 4

4. Secondary Outcome: Secondary Safety Endpoint: Number of Device-Related Serious Adverse Events
Description: Number of adjudicated device-related SAE through the 30-day visit (visit window = 30 days from procedure -5 / +15 days)
Time Frame: 30 days post procedure (-5 / +15 days)
Measure: Count of Participants; unit: Participants
Arm/Group | All Subjects
Number analyzed (Participants) | 50
Participants
  Yes | 0
  No | 46
  Withdrawn | 4

5. Secondary Outcome: Secondary Safety Endpoint: Number of Symptomatic Recurrences of PE
Description: Number of adjudicated symptomatic recurrences of pulmonary embolism through the 30-day visit (visit window = 30 days from procedure -5 / +15 days)
Time Frame: 30 days post procedure (-5 / +15 days)
Measure: Count of Participants; unit: Participants
Arm/Group | All Subjects
Number analyzed (Participants) | 50
Participants
  Yes | 0
  No | 46
  Withdrawn | 4

6. Secondary Outcome: Secondary Effectiveness Endpoint: Change in Systolic Pulmonary Arterial Pressure (mmHg)
Description: Change in systolic pulmonary arterial pressure measured via right heart catheterization at the beginning of the treatment procedure and at the end of the treatment procedure
Time Frame: Intraprocedural (at beginning and end of treatment procedure (index procedure: approximately 50 minutes))
Measure: Median (Full Range); unit: mmHg
Arm/Group | All Subjects
Number analyzed (Participants) | 50
mmHg | -8.00 [-37.0 to 17.0]

7. Secondary Outcome: Secondary Effectiveness Endpoint: Number of Patients With Adjunctive Thrombolytic Use
Description: Number of patients who received adjunctive thrombolytic medication during the index procedure
Time Frame: During Procedure (index procedure: approximately 50 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | All Subjects
Number analyzed (Participants) | 50
Participants
  Yes | 0
  No | 50

ADVERSE EVENTS:
Time Frame: All AEs were followed by the Investigator until resolution or until the 30-day follow-up visit when the patient exited the study.
Description: Collection of adverse events started after the time that the informed consent form was signed and the subject was enrolled. Adverse events were monitored throughout the study up until each patient's exit from the study.
Arm/Group | All Subjects
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 10/50
Other Adverse Events (participants affected / at risk) | 11/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=50)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 2 (2)
Vascular access site haematoma (Injury, poisoning and procedural complications) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute myocardial infarction (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Adrenal insufficiency (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=50)
Deep Vein Thrombosis (Vascular disorders) | 2 (2)
Blood Loss Anaemia (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypertensive emergency (Vascular disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
COVID-19 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Headache (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-08-11): https://cdn.clinicaltrials.gov/large-docs/63/NCT05560763/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-04): https://cdn.clinicaltrials.gov/large-docs/63/NCT05560763/SAP_001.pdf